CLINICAL TRIAL: NCT04102904
Title: A Multi-centre Validation Cohort Study Evaluating the Chemical Elements Content in Semen and Expressed Prostatic Secretions in the Diagnosis and Characterisation of Prostate Cancer, in Men Identified as Having a Risk of Prostate Cancer
Brief Title: The Prostate Liquid Study (PLiS)
Acronym: PLiS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0526
Record Dates: First submitted 2019-09-13; First posted 2019-09-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Patients will be asked to donate a semen sample which will be analysed and compared with their eventual diagnosis.

SUMMARY:
A multi-site study to evaluate the potential use of the ChEC test of seminal fluid as an additional triage test in stratifying patients for further tests.

DETAILED DESCRIPTION:
A biomarker is a molecular substance that is an indicator of a biological condition. Cambridge Oncometrix believe that a semen biomarker may be able to predict the presence of prostate cancer. This study will allow work to be carried out on semen samples donated by men who have been identified by their GPs as having a risk of prostate cancer. Normally, GPs refer men with symptoms or a raised PSA to hospital to have an MRI scan and a biopsy.

The PLiS research team at the hospital will contact potential patients, who have been referred by their GPs, before they have an MRI or a biopsy, ask them if they are willing to take part in the study, consent them and ask them to provide a semen sample. Semen samples will be produced by the potential participants at home into a seminal fluid collection container, they will also have to complete a study questionnaire. Both the sample and the questionnaire will be returned to the central laboratory in Cambridge using the stamped addressed envelope provided.

In addition to providing a semen sample and completing a questionnaire, each participant will have two blood tests to measure male hormones. Participants then exit the trial and their usual care carries on from this point. The PLiS study will register 400 men and of those it is hoped that 300 of them will be able to provide semen.

ELIGIBILITY:
Inclusion Criteria:

1. - Men over 40 years old with suspected prostate cancer who have been referred to a secondary care
2. - Men able to produce a semen sample
3. - Men able to have a prostate mpMRI
4. - Men who have given their written informed consent

Exclusion Criteria:

1. - Previous history of prostate biopsy
2. - Contraindication to MRI
3. - Previous history of prostate surgery
4. - Treatment with 5-alpha-reductase inhibitors at time of registration or during the prior 6 months
5. - Evidence of urinary tract infection or history of acute prostatitis within the last month
6. - Androgen replacement therapy within the last 3 months
7. - Any other medical condition precluding standard diagnostic workup and collection of semen samples.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men over the age of 40 who have been referred for secondary care due to suspicion of prostate cancer who are able to have an MRI scan and produce a semen sample.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Metrics of the ChEC-S test | 18 Months
  Sensitivity, specificity, negative and positive predictive values, and reciever operating characteristics (area under the curve) in the participants with a high risk of prostate cancer using mpMRI as a clinical reference standard.
Threshold | 18 Months
  Optimal threshold for the ChEC-S diagnostic score
Proportion | 18 Months
  Proportion of men who could safely avoid an MRI targeted biopsy as determined by specificity and negative predictive values of the ChEC-S test at the optimal ChEC-S test cut-off levels

SECONDARY OUTCOMES:
Proportion of significance | 18 Months
  Proportion of men correctly identified of ChEC-S test to have clinically significant prostate cancer
Value | 18 Months
  Value of the ChEC-S test as a prognostic marker of clinically significant prostate cancer (a positive predictive value). Evaluation of the prognostic power of the chemical elements as biomarkers of aggressive prostate cancer using Gleason score as clinical reference standard.
Hypogonadism Impact | 18 Months
  The impact of hypogonadism on the ChEC-S score
Resource | 18 Months
  Resource use and costs for further economic evaluation

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University College Hospital, London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich